CLINICAL TRIAL: NCT00157898
Title: A Prospective, Multicenter, Open, Randomized, Comparative Study to Evaluate the Safety and Efficacy of Ertapenem Versus it's Comparator in the Treatment of Complicated Intra-abdominal Infections in Adults
Brief Title: A Study to Evaluate Ertapenem Versus It's Comparator in the Treatment of Complicated Intra-abdominal Infections in Adults (0826-050)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0826-050; MK0826-050; 2005_068
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Complicated Intra-abdominal Infection
MeSH Terms: interventions — Ertapenem; Metronidazole

INTERVENTIONS:
Drug: MK0826; ertapenem sodium
Drug: Comparator: ceftriaxone + metronidazole

SUMMARY:
This was a prospective, randomized, controlled, open, and multi-center trial conducted to compare the clinical efficacy and safety of ertapenem with it's comparator before or following adequate surgical management of complicated intra-abdominal infection.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 75 who have complicated intra-abdominal infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-01; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Favorable clinical response at 7-14 days after treatment

SECONDARY OUTCOMES:
Favorable microbiologic response at 7-14 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html